CLINICAL TRIAL: NCT06394193
Title: Va Meh Du: An Intervention to Promote Mental Wellness Among Karenni Young Adults and Children
Brief Title: Va Meh Du Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00111733
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-04

CONDITIONS: Mental Health Wellness
Keywords: physical activity; Karenni; community support
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The 20 anticipated coach participants, 10 will be assigned to the intervention and 10 will be assigned to the comparison group; assignment will occur based on availability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community-based Participatory Research (Experimental): Coaching a six-month soccer program with the Va Meh Du intervention
  Interventions: Behavioral: Community-based participatory research intervention
- Standard Soccer Coaching (No Intervention): Standard six month soccer program without the Va Meh Du Intervention.

INTERVENTIONS:
Behavioral: Community-based participatory research intervention — Two training sessions (roughly two hours each) to train them in the intervention structure and curriculum
  Arms: Community-based Participatory Research

SUMMARY:
This study is a conceptually integrated community-based participatory research study that includes the design and evaluation of an intervention to promote mental wellness and physical activity for Karenni children and young adults.

DETAILED DESCRIPTION:
This study is a non-randomized equivalent design of an implementation and evaluation of an intervention to promote mental health and wellness among Karenni young adults and children by engaging in evidence-based mental health practices, relationship-building and physical activity through the team sport of soccer.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as Karenni
* Speaks English or Karenni
* Currently lives in Forsyth County
* Male gender
* Consents to participate

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Men/male
Enrollment: 16 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Psychological well-being | Month 6
  Flourishing Scale (FS-8). FS-8 is an eight-item validated survey measuring psychological well-being by addressing different aspects of positive mental health (e.g. I lead a purposeful and meaningful life). Participants indicate their disagreement or agreement with each statement on a 7-point Likert scale, from 1 (strongly disagree) to 7 (strongly agree). Scores range from 8 to 56, with higher scores indicating better levels of psychological well-being.

SECONDARY OUTCOMES:
Coach retention rate | Month 6
  count and percentage for coach retention
Player retention rate | Month 6
  count and percentage for player retention
Coach completion rate | Month 6
  count and percentage for coach participants, including participation in coach training and in soccer practice sessions
Player completion rate | Month 6
  player count and percentage for player participants, including participation in in soccer practice sessions

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Daniel, PhD, Principal Investigator — Wake Forest University Health Sciences; Ana Sucaldito, PhD, MPH, Principal Investigator — University of North Carolina
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-05-24): https://cdn.clinicaltrials.gov/large-docs/93/NCT06394193/ICF_000.pdf